CLINICAL TRIAL: NCT01094197
Title: Evaluation to Determine Whether Transfusion-associated Microchimerism Involves Engraftment With Hematopoietic Progenitor Cells
Brief Title: Detailed Evaluation of Microchimerism
Status: Withdrawn | Type: Observational
Why Stopped: Investigators could not identify subjects who met all inclusion criteria.
Sponsor: Vitalant Research Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 695; R01HL083388 (NIH); 1R01HL083388 (NIH)
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Chimerism; Blood Transfusion; Wounds and Injuries; Hematopoiesis
Keywords: Transfusion-associated microchimerism; Injuries; Leukocytes
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Leukapheresis filtrate and/or whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transfused microchimeric subject: Former trauma patient who underwent blood transfusion and has recent evidence of long-term transfusion-associated microchimerism

SUMMARY:
Individuals who experience traumatic injury often require blood transfusion. In some individuals who receive blood after an injury, white blood cells from a person who donated blood may remain in the body for years, a condition known as microchimerism. This study is designed to examine a group of people who are known to have long-term microchimerism and, through analysis of their blood, determine whether there is evidence that the microchimerism involves blood stem cells that can become any type of blood cell (red blood cells, white blood cells, or platelets) and that might be a permanent part of the body.

DETAILED DESCRIPTION:
Transfusion-associated microchimerism, the persistence of donor white blood cells months or years after transfusion in the recipient, has been observed in approximately 10-15% of transfused trauma patients. Previous studies suggest that the microchimeric cells include multiple immunophenotypes of leukocytes (CD4+, CD8+, CD15+, and CD19+) and that they can persist for decades, features suggestive of hematopoietic engraftment.

In this study, ten subjects known to have long-term microchimerism will undergo either leukapheresis (a blood filtering procedure) or collection of a 500 mL whole blood sample (the amount of a standard blood donation). These samples will then be analyzed to determine whether the microchimeric (donor) cells include hematopoietic stem cells (CD34+) and precursor cells in the red blood cell, white blood cell, and platelet lineages.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrated long-term microchimerism following transfusion for traumatic injury

Exclusion Criteria:

* Prior bone marrow or solid organ transplantation
* Pregnancy
* Blood transfusion within the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previous study participants
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Busch, MD, PhD, Principal Investigator — Vitalant Research Institute
Locations (1):
- University of California, Davis, Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Utter GH, Owings JT, Lee TH, Paglieroni TG, Reed WF, Gosselin RC, Holland PV, Busch MP. Blood transfusion is associated with donor leukocyte microchimerism in trauma patients. J Trauma. 2004 Oct;57(4):702-7; discussion 707-8. doi: 10.1097/01.ta.0000140666.15972.37. PMID 15514522
- [Background] Lee TH, Paglieroni T, Utter GH, Chafets D, Gosselin RC, Reed W, Owings JT, Holland PV, Busch MP. High-level long-term white blood cell microchimerism after transfusion of leukoreduced blood components to patients resuscitated after severe traumatic injury. Transfusion. 2005 Aug;45(8):1280-90. doi: 10.1111/j.1537-2995.2005.00201.x. PMID 16078913
- [Background] Utter GH, Reed WF, Lee TH, Busch MP. Transfusion-associated microchimerism. Vox Sang. 2007 Oct;93(3):188-95. doi: 10.1111/j.1423-0410.2007.00954.x. PMID 17845255
- [Background] Utter GH, Lee TH, Rivers RM, Montalvo L, Wen L, Chafets DM, Reed WF, Busch MP. Microchimerism decades after transfusion among combat-injured US veterans from the Vietnam, Korean, and World War II conflicts. Transfusion. 2008 Aug;48(8):1609-15. doi: 10.1111/j.1537-2995.2008.01758.x. Epub 2008 May 22. PMID 18503616